CLINICAL TRIAL: NCT00001586
Title: Treatment of Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL): DNA Microarray Gene Expression Analysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Wyndham Wilson, M.D., Principal investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 970178; 97-C-0178; NCT00019370 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Genetics; Bone Marrow Transplantation; Immunosuppression; T Lymphocytes; Marrow Purging
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Intermediate Risk B-Cell Pts (Experimental): Previously untreated low or intermediate risk B-cell chronic lymphocytic lymphoma (CLL)/small lymphocytic lymphoma (SLL) patients (pts) not requiring chemotherapy. No rituximab fludarabine administered. Eligible to donate cells.
  Interventions: Other: Leukemic or stroma cells
- Intermediate-high Risk B-Cell Pts (Experimental): Previously untreated intermediate or high risk B-cell chronic lymphocytic lymphoma (CLL)/small lymphocytic lymphoma (SLL) patients requiring chemotherapy. Rituximab 375 mg/m^2 by infusion on day 1, cycle 1 followed by fludarabine on day 2-6, 25 mg/m^2 day x 5 days administered as an intravenous push or intravenous piggyback over 10-30 minutes, repeated every 28 days.
  Interventions: Biological: Rituximab; Drug: Fludarabine phosphate

INTERVENTIONS:
Biological: Rituximab — Rituxan
  Other Names: Rituximab 375 mg/m^2 by infusion on day 1, cycle 1. Repeated every 28 days.
  Arms: Intermediate-high Risk B-Cell Pts
Drug: Fludarabine phosphate — Fludara
  Other Names: Fludarabine on day 2-6, 25 mg/m^2 day x 5 days administered as an intravenous push or intravenous piggyback over 10-30 minutes, repeated every 28 days.
  Arms: Intermediate-high Risk B-Cell Pts
Other: Leukemic or stroma cells — Patients are eligible to donate cells for the purpose of analyzing leukemic cells. Cells can be donated by apheresis (e.g. 60-90 minute intravenous technique), lymph node biopsy (e.g. 3 biopsy/excision of lymph nodes)bone marrow biopsy (e.g. 2-4 separate bone marrow biopsies), and bone marrow aspiration (e.g. 3 to 5cc of marrow per aspirate).
  Arms: Low-Intermediate Risk B-Cell Pts

SUMMARY:
Background:

* Combined therapy with rituximab and fludarabine is the treatment of choice for advanced stage chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL).
* A new technology called deoxyribonucleic acid (DNA) microarray can be used to gain knowledge about the genetic basis of CLL/SLL.
* Genetic studies of CLL/SLL may improve our understanding of what happens in the disease, help determine which patients are most likely to respond to treatment with fludarabine and rituximab, and identify new treatments.

Objectives:

-To gain further knowledge about CLL/SLL and the role of rituximab and fludarabine in treating the disease.

Eligibility:

-Patients 18 years of age and older with low, intermediate or high-risk CLL/SLL.

Design:

* Patients with low-risk CLL/SLL do not receive treatment, but are followed every 3 to 6 months and donate cells (through apheresis) or lymph nodes, or both, for research purposes.
* Patients with intermediate or high-risk CLL/SLL receive standard treatment with rituximab and fludarabine for six 28-day treatment cycles. Rituximab is given on day 1 and fludarabine is given on days 1-5. (For the first cycle only, fludarabine treatment starts on day 2. This delay permits blood sampling on day 1 for the effect of rituximab on white blood cells.)
* Laboratory tests and imaging studies are done periodically to monitor drug side effects and the response to treatment. Tests include bone marrow biopsy and aspiration, blood tests and x-rays, including positron emission tomography (PET) and computed tomography (CT) scans.

DETAILED DESCRIPTION:
Background:

* Due to their synergistic action and non-overlapping toxicity profiles, the combination of Rituximab and Fludarabine is the treatment of choice for advanced stage chronic lymphocytic lymphoma (CLL)/small lymphocytic lymphoma (SLL).
* As such, we have designed this protocol to better understand the genetic basis of CLL/SLL, to identify predictors of treatment response and to study the molecular effects of Rituximab Fludarabine on the leukemic cells.
* A new technology utilizing complementary deoxyribonucleic acid (cDNA) microarrays now permits the simultaneous quantitation of the expression of thousands of genes; this methodology can evaluate defined cellular pathways, and also discover novel genes influencing cell biology.
* In addition to improving our understanding of the pathogenesis of CLL/SLL, these molecular studies may identify new therapeutic targets in CLL/SLL, and may help to identify those CLL/SLL patients most likely to respond to the combination of Fludarabine and Rituximab.

Objectives:

* Evaluate CLL/SLL patients during and following Rituximab Fludarabine chemotherapy for changes in lymphocyte gene expression using DNA microarray analysis.
* Evaluate gene expression by DNA microarray analysis of leukemic cells in blood, bone marrow and lymph nodes.

Eligibility:

* Low, Intermediate or High-Risk Category of CLL/SLL, using the Modified Three- Stage Rai Staging System
* Age greater than or equal to 18 years.
* Patients must have received no previous cytotoxic or monoclonal antibody therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Patients must not be pregnant or breast-feeding.
* Patients with active autoimmune hemolytic anemia (AIHA)) grade III or higher (transfusion or steroids indicated) or immune thrombocytopenia (ITP) grade III or higher (platelets less than 50,000/microL) shall not be enrolled.
* Any patient with a medical condition that requires chronic use of corticosteroids shall not be enrolled.

Design:

* Patients who do not require treatment will be followed every 3-6 months and will donate cellular products, bone marrow biopsies, bone marrow aspirates and/or lymph nodes for research purposes.
* Patients who do require treatment will received the standard dose of the Rituximab monoclonal antibody and the standard dose of Fludarabine for a total of six cycles. In the first cycle, Rituximab will be given on day 1 with Fludarabine being given on days 2-6. This will allow for appropriate samplings of the effects of Rituximab on lymphocytes before during and at the end of the first 24 hours. In subsequent cycles 2-6, the Rituximab and day 1 Fludarabine can both be given on day 1.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of chronic lymphocytic lymphoma (CLL)/small lymphocytic lymphoma (SLL) will be made according to the World Health Organization (WHO) diagnostic classification. A lymphocyte count in excess of 5000/mcl is typically found in the leukemic variant but is not a pre-requisite for a diagnosis of SLL. Low, Intermediate or High-Risk Category of CLL/SLL, using the Modified Three-Stage Rai Staging System as follows:

Risk Category: Low Risk

Rai Stage: 0

Clinical Features: Elevated blood and marrow lymphocyte numbers only (L). (lymphocytes greater than 5000/microl in blood, and lymphocytes greater than 30 percent in marrow).

Risk Category: Intermediate Risk

Rai Stage: I

Clinical Features: L + enlarged lymph nodes (LN)

Risk Category: Intermediate Risk

Rai Stage: II

Clinical Features: L + enlarged spleen or liver

Risk Category: High Risk

Rai Stage: III

Clinical Features: L + anemia (Hemoglobin less than 11 gm/dl)

Risk Category: High Risk

Rai Stage: IV

Clinical Features: L + thrombocytopenia (platelets less than 100,000/microl)

Patients in the modified Rai high risk group and select patients in the intermediate risk group will undergo treatment with Rituximab Fludarabine. To meet treatment criteria patients in the intermediate risk group should have evidence of active disease as demonstrated by at least one of the following criteria:

1. massive or progressive splenomegaly or lymphadenopathy;
2. presence of weight loss greater than 10% over the preceding 6 months;
3. constitutional symptoms of extreme fatigue, night sweats or recurrent fever of greater than 100 degrees F (documented fevers must be occurring without evidence of specific infection), and bone pain;
4. progressive lymphocytosis with an increase of greater than 50% over a 2 month period, or an anticipated doubling time of less than 6 months;
5. chronic infections either increased number or prolonged infections;
6. other high risk prognostic indicators such as excess elevation of beta-2-microglobulin, cluster differentiation 38 (CD38) expression and adverse cytogenetics may be used to better appraise the risk in each individual patient.

Patients with a diagnosis of CLL/SLL who do not meet the eligibility criteria for receiving Rituximab and Fludarabine (are not intermediate- or high-risk CLL/SLL), can enroll on the protocol for the purpose of donating cellular products. Such patients will not receive rituximab and fludarabine chemotherapy. At a later date, if it is documented that the patient does meet the criteria, then the patient may receive Rituximab and Fludarabine (after discussion with the Principal Investigator).

In a limited number of cases, patients with low-risk CLL/SLL may be initiated on Rituximab and Fludarabine treatment. For example, individuals who are candidates for bone marrow transplantation may be started on Rituximab Fludarabine as an induction regimen prior to transplantation. Additionally, some low-risk patients may be started on Rituximab and Fludarabine for psychological reasons (patient insistence on starting chemotherapy prior to disease progression). However, it must be stressed that low-risk CLL/SLL patients will be discouraged from initiating therapy except in these specific cases.

Age greater than or equal to 18 years of age.

Patients must have received no prior cytotoxic or monoclonal antibody therapy.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

Required initial laboratory tests: Blood urea nitrogen (BUN) and Creatinine values must be less than or equal to 1.5 times the normal values; alternatively, patients with creatinine clearance of greater than 50 ml per minute will also be eligible. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) values must be less than or equal to 2.0 times normal values; patients with laboratory values greater than these levels may be enrolled on the protocol (after a specific approval from the Principal Investigator) if the values are due to a known, pre-existing liver disease. Bilirubin must be less than or equal to 2.0 mg/dl unless due to Gilbert's disease.

The patient must be competent to sign an informed consent, and sign the protocol consent form.

EXCLUSION CRITERIA:

Patients must not be pregnant or breastfeeding.

Patients with active autoimmune hemolytic anemia (AIHA)) grade III or higher (transfusion or steroids indicated) or immune thrombocytopenia (ITP) grade III or higher (platelets less than 50,000/microL) shall not be enrolled. Patients with a history of prior therapy to control either AIHA or ITP will be eligible, provided they do not require maintenance corticosteroids, and have not received monoclonal antibody therapy in the past 6 months. Patients developing AIHA or ITP on protocol may be managed as medically indicated on protocol but will generally not undergo fludarabine/rituximab treatment until resolution of hemolysis or thrombocytopenia to less than grade III.

Any patient with a medical condition that requires chronic use of corticosteroids shall not be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 1997-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H Wilson, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rai KR, Sawitsky A, Cronkite EP, Chanana AD, Levy RN, Pasternack BS. Clinical staging of chronic lymphocytic leukemia. Blood. 1975 Aug;46(2):219-34. PMID 1139039
- [Background] Keating MJ. Fludarabine phosphate in the treatment of chronic lymphocytic leukemia. Semin Oncol. 1990 Oct;17(5 Suppl 8):49-62. PMID 1699283
- [Background] Raife TJ, Demetroulis EM, Lentz SR. Regulation of thrombomodulin expression by all-trans retinoic acid and tumor necrosis factor-alpha: differential responses in keratinocytes and endothelial cells. Blood. 1996 Sep 15;88(6):2043-9. PMID 8822923
- [Derived] Mo CC, Njuguna N, Beum PV, Lindorfer MA, Vire B, Lee E, Marti G, Wilson WH, Taylor RP, Wiestner A. Rapid clearance of rituximab may contribute to the continued high incidence of autoimmune hematologic complications of chemoimmunotherapy for chronic lymphocytic leukemia. Haematologica. 2013 Aug;98(8):1259-63. doi: 10.3324/haematol.2012.080929. Epub 2013 May 28. PMID 23716541
- [Derived] Herishanu Y, Perez-Galan P, Liu D, Biancotto A, Pittaluga S, Vire B, Gibellini F, Njuguna N, Lee E, Stennett L, Raghavachari N, Liu P, McCoy JP, Raffeld M, Stetler-Stevenson M, Yuan C, Sherry R, Arthur DC, Maric I, White T, Marti GE, Munson P, Wilson WH, Wiestner A. The lymph node microenvironment promotes B-cell receptor signaling, NF-kappaB activation, and tumor proliferation in chronic lymphocytic leukemia. Blood. 2011 Jan 13;117(2):563-74. doi: 10.1182/blood-2010-05-284984. Epub 2010 Oct 12. PMID 20940416
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1997-C-0178.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intermediate-high Risk B-Cell Pts | Low-Intermediate Risk B-Cell Pts
Started | 49 | 56
Completed | 49 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low-Intermediate Risk B-Cell Pts: Previously untreated low or intermediate risk B-cell chronic lymphocytic lymphoma (CLL)/small lymphocytic lymphoma (SLL) patients (pts) not requiring chemotherapy. No rituximab fludarabine administered.
- Total: Total of all reporting groups
Arm/Group | Intermediate-high Risk B-Cell Pts | Low-Intermediate Risk B-Cell Pts | Total
Number analyzed (Participants) | 49 | 56 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 78
  >=65 years | 10 | 17 | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 56.2 (9.34) | 58.42 (11.32) | 57.98 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 30 | 35 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 49 | 55 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 42 | 52 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 49 | 56 | 105

OUTCOME MEASURES:

1. Primary Outcome: Change in Gene Expression Post Chemo
Description: Changes in lymphocyte gene expression was measured by deoxyribonucleic acid (DNA) microarray analysis of circulating leukemic cells after completion of study treatment. A change in expression is defined as a >50% increase in circulating leukemic cells or a 30% decrease in circulating leukemic cells.
Time Frame: 6 hours post treatment, and 24 hours post treatment
Population: There were only 12 patients analyzed for various reasons such as timing of treatment, ability to collect samples, and viability of samples.
Measure: Number; unit: Percent change in cells
Arm/Group | Intermediate-high Risk B-Cell Pts | Low-Intermediate Risk B-Cell Pts
Number analyzed (Participants) | 12 | 0
Percent change in cells
  6 hours post treatment (e.g. ># cells) | 30 |
  24 hours post treatment (e.g. > # cells) | 50 |

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 13 years, 10.5 months
Population: The low-intermediate risk patients received no treatment so their tissue/blood was not analyzed for change.
Measure: Number; unit: Participants
Arm/Group | Intermediate-high Risk B-Cell Pts | Low-Intermediate Risk B-Cell Pts
Number analyzed (Participants) | 49 | 0
Participants | 18 |

ADVERSE EVENTS:
Description: The low-intermediate risk B cell patients did not receive any treatment. No adverse events were collected for these patients. This group does not have adverse events.
Arm/Group | Intermediate-high Risk B-Cell Pts | Low-Intermediate Risk B-Cell Pts
Serious Adverse Events (participants affected / at risk) | 19/49 | 0/0
Other Adverse Events (participants affected / at risk) | 18/49 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermediate-high Risk B-Cell Pts (N=49) | Low-Intermediate Risk B-Cell Pts (N=0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (3) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 0 (0)
Autoimmune reaction (Immune system disorders) | 4 (4) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 8 (11) | 0 (0)
Hemorrhage, GI::Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC < 1.0 x 10e9/L)::Anal/perianal
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::External ear (otitis externa) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 1 (1) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 19 (31) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 18 (36) | 0 (0)
Pain::Neuralgia/peripheral nerve (Nervous system disorders) | 1 (1) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermediate-high Risk B-Cell Pts (N=49) | Low-Intermediate Risk B-Cell Pts (N=0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 10 (11) | 0 (0)
Rhinorrhea (Immune system disorders) | 15 (25) | 0 (0)
Alkaline phosphatase (Hepatobiliary disorders) | 3 (3) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3 (4) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 5 (6) | 0 (0)
Anorexia (Gastrointestinal disorders) | 6 (6) | 0 (0)
Autoimmune reaction (Immune system disorders) | 3 (3) | 0 (0)
Bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 4 (6) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Cardiac arrhythmia - Other, Specify, unknown (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Creatinine (Renal and urinary disorders) | 1 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Edema: limb (General disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (5) | 0 (0)
Febrile neutropenia (Infections and infestations) | 3 (3) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 8 (9) | 0 (0)
Glucose, serum-low (hyperglycemia) (Metabolism and nutrition disorders) | 12 (17) | 0 (0)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Oral cavity (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory: Nose (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Transfusion (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Infection w/neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Hemoptysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper aerodigestive NOS (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 2 (2) | 0 (0)
Infection with unknown ANC::Skin (cellulites) (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 2 (2) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 16 (55) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 13 (29) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Mood alteration::Anxiety (Nervous system disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (16) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 18 (55) | 0 (0)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pain::Abdomen NOS (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Pain::Chest wall (Cardiac disorders) | 1 (1) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 18 (45) | 0 (0)
Bone pain (General disorders) | 4 (6) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No